CLINICAL TRIAL: NCT04502732
Title: Direct Comparison of Short- And Long-Term Gastric Emptying By Nuclear Scintigraphy and Gastric Emptying Breath Test in Subjects Undergoing Endoscopic Gastric Remodeling For Weight Loss
Brief Title: Gastric Emptying Using Two Imaging Methods for Those Who Have Undergone POSE2 Weight Loss Procedure
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit sufficient participants form parent study following protocol expansion
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barham K. Abu Dayyeh, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 20-002882
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: NSSM and GEBT
  Interventions: Other: NSSM and GEBT

INTERVENTIONS:
Other: NSSM and GEBT — The time to half gastric emptying (T1/2) will be assessed via Gastric Emptying Breath Tests (GEBT) and Nuclear Scintigraphy of a Solid Meal (NSSM) at baseline, 2 months, and 6 months. This data will be collected from seven adult subjects, with obesity, who have recently received Endoscopic Bariatric and Metabolic Therapy.

SUMMARY:
The purpose of this study is to compare a less invasive breath test against the current standard for assessing gastric (stomach) emptying. The current standard of care is a procedure called Nuclear Scintigraphy of a Solid Meal (NSSM). This study will compare this method to a Gastric Emptying Breath Test (GEBT).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 22-65 years of age at time of enrollment
* Subjects must already be consented to 17-007934 or 19-001254
* Subject must be agreeable and compliant with study requirements, including up to three (baseline, 2 month, and 6 month) visits, as well as undergoing GEBT and NSSM testing.
* If female, must be post-menopausal, surgically sterile, or agree to practice a form of birth control or abstinence during year of study and have negative serum HCG at screening/baseline
* Must be willing and able to travel, as needed, to the Investigator's office to complete all routine follow-up visits

Exclusion Criteria:

* Persons presently or soon to be incarcerated
* Females who are pregnant or suspect they may be pregnant
* Persons with nicotine and/or alcohol dependence
* Patients with cognitive impairment that limits their ability to make autonomous decisions
* Known allergies or sensitivities to study materials (eggs and spirulina)
* Assessed, by the physician or delegate, that enrollment would not be appropriate

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those eligible from relevant sub-studies.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Change of T1/2 | Baseline, 2 months, 6 months
  The aim of this study is to compare baseline, early post-procedural (2 month), and delayed post-procedural (6 month) T1/2, as assessed by both GEBT and NSSM, in seven adult subjects with obesity who have underwent an EGRWL procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Barham Abu Dayyeh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials